CLINICAL TRIAL: NCT02367378
Title: Minimally Invasive Surgery for Spine Metastases - A Prospective Study
Brief Title: Minimally Invasive Surgery (MIS) for Spine Metastases
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 12-0161
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Spine Metastases
Keywords: Minimally invasive surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MIS: Those who received minimally invasive surgical procedures
- Control: Those who received treatments which include surgical resection, chemotherapy, and radiotherapy.

SUMMARY:
The purpose of this study is to collect information on the effect of minimally invasive spine tumor decompression on treated patients. This treatment option is less invasive that the standard surgical decompression and is expected to result in better wound healing, decreased tissue trauma, and decreased pain after surgery.

DETAILED DESCRIPTION:
This is a prospective study designed to analyze the impact that minimally invasive spine tumor decompression has upon quality of life, neurological morbidity, pain, and mortality. Prospective findings will be compared with historical controls to determine whether the minimally invasive approach offers better outcomes than traditional treatment methods.

ELIGIBILITY:
Inclusion Criteria:

* undergone minimally invasive surgery
* over 18 years of age

Exclusion Criteria:

* unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chart review of patients having undergone minimally invasive surgery of spine metastases, 18 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06-13 (Actual); Study Completion 2016-06-13 (Actual)

PRIMARY OUTCOMES:
Survival time | up to 2 years
  Survival time in days

SECONDARY OUTCOMES:
Ambulation Index | up to 2 years
  Hauser Ambulation Index to assess mobility by evaluating the time and degree of assistance required to walk 25 feet. Scores range from 0 (asymptomatic and fully active) to 10 (bedridden).
Cobb Angle | up to 2 years
  The Cobb angle is used to quantify the magnitude of spinal deformities.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Jenkins, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States